CLINICAL TRIAL: NCT05313100
Title: The Evaluation of the Effects of the Use of Rocuronium and Sugammadex on Neuromuscular Block in Smoker
Brief Title: Sugammadex and Smoker's Neuromuscular Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2012.04.HD.067
Record Dates: First submitted 2015-08-06; First posted 2022-04-06 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Neuromuscular Blockade; Smoking
Keywords: sugammadex; smoking; neuromuscular blockade
MeSH Terms: conditions — Smoking | interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smokers (Active Comparator): The patients who have smoked at least 10 packs or have been smoking for 10 years and currently smoking were included in the smoker group At the end of operation for reversal of neuromuscular blockade sugammadex used.
  Interventions: Drug: sugammadex
- Nonsmokers (Sham Comparator): The patients who never smoked were included in the non-smoker group At the end of operation for reversal of neuromuscular blockade sugammadex used.
  Interventions: Drug: sugammadex

INTERVENTIONS:
Drug: sugammadex — At the end of the operation, at least 15 minutes after the last dose of rocuronium, sugammadex 2 mg / kg was administered both of groups
  Other Names: bridion

SUMMARY:
We compared the durations of antagonizing and of the severity of effect of sugammadex used in antagonizing the rocuronium in smoker and non-smoker total 40 patients with using Train of Four(TOF) neuromuscular monitorization.

DETAILED DESCRIPTION:
40 patients from American Society of Anesthesiologist (ASA) I- II class, being smokers for at least 10 years or non-smokers, who will undergo elective surgery were included in this randomized prospective study. Patients underwent routine monitoring and neuromuscular monitoring. Propofol 2 mg/kg and intravenous fentanyl 1 mcg/kg were applied at induction. After the loss of eyelash reflex, intravenous rocuronium 0,6 mg/kg was administered. The patient was intubated at a Train of Four count of 2. Anesthesia was continued with 50% O2 + 50% air and sevoflurane 2 % . Rocuronium 0,15 mg/kg was administered when TOF (Train of Four) counter reached 2 during the operation. Sugammadex 2 mg/kg was administered at the end of the operation. The time to reach Train of Four values of 0,7-0,8-0,9 were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery,
* 1-2 according to the ASA ( American Society of Anesthesiologist ) physical status classification.
* Patients who have smoked at least 10 packs or have been smoking for 10 years and currently smoking
* Or never smoked patients

Exclusion Criteria:

* neuromuscular diseases
* radiotherapy and/or chemotherapy anamnesis,
* liver and/or renal disease,
* electrolyte balance,
* history of drug use which affects neuromuscular transmission,
* Body Mass Index (BMI) of more than 27,
* use alcohol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Neuromuscular block recovery time | six months
  Time to reach TOF %90 measurement after given neuromuscular blocker reverse agent

CONTACTS AND LOCATIONS:
Overall Officials: Gulbin Sezen, Study Director — Duzce University

IPD SHARING:
Plan to Share IPD: No